CLINICAL TRIAL: NCT02200770
Title: A Double-masked, Placebo-controlled Study With Open-label Period to Evaluate the Efficacy and Safety of MEDI-551 in Adult Subjects With Neuromyelitis Optica and Neuromyelitis Optica Spectrum Disorders.
Brief Title: N-MOmentum: A Clinical Research Study of Inebilizumab in Neuromyelitis Optica Spectrum Disorders
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CD-IA-MEDI-551-1155; 2014-000253-36 (EudraCT Number)
Record Dates: First submitted 2014-07-16; First posted 2014-07-25 (Estimated); Results first posted 2019-12-26 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Neuromyelitis Optica and Neuromyelitis Optica Spectrum Disorders
Keywords: NMO, NMOSD, Neuromyelitis Optica, Neuromyelitis Optica Spectrum Disorders, autoimmune, demyelination, MEDI-551, monoclonal antibody, Devic's syndrome, B-cell
MeSH Terms: conditions — Neuromyelitis Optica; Demyelinating Diseases | interventions — inebilizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo/Inebilizumab (Placebo Comparator): Aquaporin-4-antibody (AQP4-IgG) sero positive and sero negative participants will receive IV dose of placebo matched to inebilizumab on Day 1 and Day 15 of the RCP. The participants who enter OLP will receive IV inebilizumab 300 mg on both Day 1 and Day 15, followed by a single IV dose of inebilizumab 300 mg every 6 months until maximum of 3 years after the last participant enters the OLP. Participants will have choice to enter in the SFP at any point during RCP or OLP and will be free to pursue other treatment options otherwise prohibited during the RCP and OLP. Participants will continue in the SFP for 12 months from last dose of study drug.
  Interventions: Drug: Inebilizumab; Other: Placebo
- Inebilizumab/Inebilizumab (Experimental): AQP4-IgG sero positive and sero negative participants will IV dose of inebilizumab 300 mg on Day 1 and Day 15 of RCP. The participants who enter OLP will receive IV inebilizumab 300 mg on Day 1 and matching placebo on Day 15, followed by a single IV dose of inebilizumab 300 mg every 6 months until maximum of 3 years after the last participant enters the OLP. Participants will have choice to enter in the SFP at any point during RCP or OLP and will be free to pursue other treatment options otherwise prohibited during the RCP and OLP. Participants will continue in the SFP for 12 months from last dose of study drug.
  Interventions: Drug: Inebilizumab; Other: Placebo

INTERVENTIONS:
Drug: Inebilizumab — Participants will receive IV inebilizumab 300 mg.
  Other Names: MEDI-551
Other: Placebo — Participants will receive IV placebo matched to inebilizumab.

SUMMARY:
To compare the efficacy of inebilizumab (MEDI-551) versus placebo in reducing the risk of an neuromyelitis optica/neuromyelitis optica- spectrum disorders (NMO/NMOSD) attack in participants with NMO/NMOSD.

DETAILED DESCRIPTION:
Inebilizumab is a genetically engineered humanized monoclonal antibody that binds to the B cell specific surface antigen cluster of differentiation (CD19) resulting in the depletion of B cells. Inebilizumab depletes antibody-secreting plasmablasts and some plasma cells, which are generally CD19 positive and CD20 negative.

The main objective of this study is to determine whether inebilizumab compare to placebo decreases the risk of an attack in participants with NMO/NMOSD.

This is a multicenter, multinational, randomized, double-masked, placebo controlled study with an open-label extension period to evaluate the efficacy and safety of intravenous (IV) inebilizumab in adult participants with NMO/NMOSD. After a screening period, eligible participants will enter a randomized-controlled period (RCP) of maximum 197 days where they will be randomized in a 3:1 ratio to receive either IV inebilizumab or placebo. NMO/NMOSD attacks will be evaluated by the investigator and confirmed against the attack criteria by an independent Adjudication Committee (AC). Participants for whom the attack was confirmed by the AC will be given the option to enroll into an open label period (OLP) with inebilizumab treatment. Participants who complete the RCP without experiencing an attack will be given the option to enroll into an OLP with inebilizumab treatment. The OLP will continue for a minimum of 1 year and a maximum of 3 years after the last participant enter the OLP. All participants who discontinue from the RCP or the OLP will continue in a Safety Follow-up for a total of 12 months from last dose to evaluate the long-term safety of the investigational product.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18 years or older with diagnosis of NMO/NMOSD
2. Confirmation of NMO/NMOSD status:

   1. AQP4-IgG sero-positive NMO/NMOSD with at least one attack requiring rescue therapy in the last year or two attacks requiring rescue therapy in the last 2 years
   2. AQP4-IgG sero-negative NMO with at least one attack requiring rescue therapy in the last year or two attacks requiring rescue therapy in the last 2 years
3. Able and willing to give written informed consent and comply with the requirements of the study protocol.
4. EDSS <= 7.5 (8 in special circumstances)
5. Men and women of reproductive potential must agree to use a highly effective method of birth control from screening to 6 months after final dose of the investigational product.

Exclusion Criteria:

1. Lactating and pregnant females
2. Treatment with any investigational agent within 4 weeks of screening
3. Known history of a severe allergy or reaction to any component of the investigational product formulation or history of anaphylaxis following any biologic therapy.
4. Known active severe bacterial, viral, or other infection or any major episode of infection requiring hospitalization.
5. History of alcohol, drug, or chemical abuse, or a recent history of such abuse < 1 year prior to randomization
6. Receipt of the following at any time prior to randomization:

   1. Alemtuzumab
   2. Total lymphoid irradiation
   3. Bone marrow transplant
   4. T-cell vaccination therapy
7. Receipt of rituximab or any experimental B-cell depleting agent within 6 months prior screening and B-cells below the lower limit of normal.
8. Receipt of intravenous immunoglobulin (IVIG) within 1 month prior to randomization.
9. Receipt of any of the following within 3 months prior to randomization:

   1. Natalizumab (Tysabri®).
   2. Cyclosporin
   3. Methotrexate
   4. Mitoxantrone
   5. Cyclophosphamide
   6. Tocilizumab
   7. Eculizumab
10. History of Hepatitis B and/or Hepatitis C (Hep B/C at screening)
11. Known history of a primary immunodeficiency (congenital or acquired) or an underlying condition such as human immunodeficiency virus (HIV) infection
12. History of malignancies, apart from squamous cell or basal cell carcinoma of the skin treated with documented success of curative therapy > 3 months prior to randomization
13. Any concomitant disease other than NMO/NMOSD that required treatment with oral or intravenous steroids at doses over 20 mg a day for over 21 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2020-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune, LLC MedImmune, LLC, Study Director — MedImmune LLC
Locations (87):
- United States (19):
  - Research Site, Birmingham, Alabama
  - Research Site, Sacramento, California
  - Research Site, San Francisco, California
  - Research Site, Aurora, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Maitland, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Kansas City, Kansas
  - Research Site, Baltimore, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Raleigh, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Mansfield, Ohio
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Richmond, Virginia
- Research Site, Melbourne, Australia
- Bulgaria (2):
  - Research Site, Sofia
  - Research Site, Varna
- Research Site, Vancouver, British Columbia, Canada
- Colombia (3):
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Cali
- Czechia (3):
  - Research Site, Olomouc
  - Research Site, Prague
  - Research Site, Teplice
- Estonia (2):
  - Research Site, Tallinn
  - Research Site, Tartu
- Germany (6):
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Leipzig
  - Research Site, Münster
  - Research Site, Rostock
- Research Site, Hong Kong, Hong Kong
- Hungary (3):
  - Research Site, Esztergom
  - Research Site, Nyíregyháza
  - Research Site, Szeged
- Israel (3):
  - Research Site, Jerusalem
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Japan (6):
  - Research Site, Aomori
  - Research Site, Bunkyō City
  - Research Site, Kyoto
  - Research Site, Ōta-ku
  - Research Site, Sendai
  - Research Site, Tsukuba
- Mexico (3):
  - Research Site, Mexico City
  - Research Site, Monterrey
  - Research Site, San Luis Potosí City
- Research Site, Chisinau, Moldova
- Research Site, Auckland, New Zealand
- Peru (2):
  - Research Site, Bellavista
  - Research Site, Lima
- Poland (6):
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lódz
  - Research Site, Lublin
  - Research Site, Olsztyn
  - Research Site, Warsaw
- Russia (10):
  - Research Site, Belgorod
  - Research Site, Kazan'
  - Research Site, Khabarovsk
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Saint Petersburg
  - Research Site, Ufa
- Research Site, Belgrade, Serbia
- Research Site, Cape Town, South Africa
- South Korea (3):
  - Research Site, Goyang
  - Research Site, Jongno-gu
  - Research Site, Seoul
- Research Site, Madrid, Spain
- Taiwan (3):
  - Research Site, Changhua
  - Research Site, Hualien City
  - Research Site, Tainan
- Thailand (2):
  - Research Site, Bangkok
  - Research Site, Muang
- Turkey (Türkiye) (3):
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Samsun

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Cree BAC, Kim HJ, Weinshenker BG, Pittock SJ, Wingerchuk DM, Fujihara K, Paul F, Cutter GR, Marignier R, Green AJ, Aktas O, Hartung HP, She D, Rees W, Smith M, Cimbora D, Katz E, Bennett JL; N-MOmentum study investigators. Safety and efficacy of inebilizumab for the treatment of neuromyelitis optica spectrum disorder: end-of-study results from the open-label period of the N-MOmentum trial. Lancet Neurol. 2024 Jun;23(6):588-602. doi: 10.1016/S1474-4422(24)00077-2. PMID 38760098
- [Derived] Aktas O, Hartung HP, Smith MA, Rees WA, Fujihara K, Paul F, Marignier R, Bennett JL, Kim HJ, Weinshenker BG, Pittock SJ, Wingerchuk DM, Cutter G, She D, Gunsior M, Cimbora D, Katz E, Cree BA; N-MOmentum study investigators. Serum neurofilament light chain levels at attack predict post-attack disability worsening and are mitigated by inebilizumab: analysis of four potential biomarkers in neuromyelitis optica spectrum disorder. J Neurol Neurosurg Psychiatry. 2023 Sep;94(9):757-768. doi: 10.1136/jnnp-2022-330412. Epub 2023 May 23. PMID 37221052
- [Derived] Bennett JL, Aktas O, Rees WA, Smith MA, Gunsior M, Yan L, She D, Cimbora D, Pittock SJ, Weinshenker BG, Paul F, Marignier R, Wingerchuk D, Cutter G, Green A, Hartung HP, Kim HJ, Fujihara K, Levy M, Katz E, Cree BAC; N-MOmentum study investigators. Association between B-cell depletion and attack risk in neuromyelitis optica spectrum disorder: An exploratory analysis from N-MOmentum, a double-blind, randomised, placebo-controlled, multicentre phase 2/3 trial. EBioMedicine. 2022 Dec;86:104321. doi: 10.1016/j.ebiom.2022.104321. Epub 2022 Nov 10. PMID 36370634
- [Derived] Flanagan EP, Levy M, Katz E, Cimbora D, Drappa J, Mealy MA, She D, Cree BAC. Inebilizumab for treatment of neuromyelitis optica spectrum disorder in patients with prior rituximab use from the N-MOmentum Study. Mult Scler Relat Disord. 2022 Jan;57:103352. doi: 10.1016/j.msard.2021.103352. Epub 2021 Oct 26. PMID 35158461
- [Derived] Marignier R, Bennett JL, Kim HJ, Weinshenker BG, Pittock SJ, Wingerchuk D, Fujihara K, Paul F, Cutter GR, Green AJ, Aktas O, Hartung HP, Lublin FD, Williams IM, Drappa J, She D, Cimbora D, Rees W, Smith M, Ratchford JN, Katz E, Cree BAC; N-MOmentum Study Investigators. Disability Outcomes in the N-MOmentum Trial of Inebilizumab in Neuromyelitis Optica Spectrum Disorder. Neurol Neuroimmunol Neuroinflamm. 2021 Mar 26;8(3):e978. doi: 10.1212/NXI.0000000000000978. Print 2021 May. PMID 33771837
- [Derived] Aktas O, Smith MA, Rees WA, Bennett JL, She D, Katz E, Cree BAC; N-MOmentum scientific group and the N-MOmentum study investigators. Serum Glial Fibrillary Acidic Protein: A Neuromyelitis Optica Spectrum Disorder Biomarker. Ann Neurol. 2021 May;89(5):895-910. doi: 10.1002/ana.26067. Epub 2021 Mar 30. PMID 33724534
- [Derived] Cree BA, Bennett JL, Kim HJ, Weinshenker BG, Pittock SJ, Wingerchuk D, Fujihara K, Paul F, Cutter GR, Marignier R, Green AJ, Aktas O, Hartung HP, Williams IM, Drappa J, She D, Cimbora D, Rees W, Ratchford JN, Katz E. Sensitivity analysis of the primary endpoint from the N-MOmentum study of inebilizumab in NMOSD. Mult Scler. 2021 Nov;27(13):2052-2061. doi: 10.1177/1352458521988926. Epub 2021 Feb 4. PMID 33538237
- [Derived] Cree BAC, Bennett JL, Kim HJ, Weinshenker BG, Pittock SJ, Wingerchuk DM, Fujihara K, Paul F, Cutter GR, Marignier R, Green AJ, Aktas O, Hartung HP, Lublin FD, Drappa J, Barron G, Madani S, Ratchford JN, She D, Cimbora D, Katz E; N-MOmentum study investigators. Inebilizumab for the treatment of neuromyelitis optica spectrum disorder (N-MOmentum): a double-blind, randomised placebo-controlled phase 2/3 trial. Lancet. 2019 Oct 12;394(10206):1352-1363. doi: 10.1016/S0140-6736(19)31817-3. Epub 2019 Sep 5. PMID 31495497
- [Derived] Cree BA, Bennett JL, Sheehan M, Cohen J, Hartung HP, Aktas O, Kim HJ, Paul F, Pittock S, Weinshenker B, Wingerchuk D, Fujihara K, Cutter G, Patra K, Flor A, Barron G, Madani S, Ratchford JN, Katz E. Placebo-controlled study in neuromyelitis optica-Ethical and design considerations. Mult Scler. 2016 Jun;22(7):862-72. doi: 10.1177/1352458515620934. Epub 2015 Dec 14. PMID 26666258
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=CD-IA-MEDI-551-1155&attachmentIdentifier=ae7e7dac-afeb-4a4e-bf68-5ce2e36292b8&fileName=statistical_analysis_plan_cd-ia-medi-551-1155_amendment_4-redacted_PDFA.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo/Inebilizumab: Aquaporin-4-antibody (AQP4-IgG) sero positive and sero negative participants received IV dose of placebo matched to inebilizumab on Day 1 and Day 15 of the RCP. The participants who entered OLP received IV inebilizumab 300 mg on both Day 1 and Day 15, followed by a single IV dose of inebilizumab 300 mg every 6 months until maximum of 3 years after the last participant enters the OLP. Participants had choice to enter in the SFP at any point during RCP or OLP and were free to pursue other treatment options otherwise prohibited during the RCP and OLP. Participants continued in the SFP for 12 months from last dose of study drug.
- Inebilizumab/Inebilizumab: AQP4-IgG sero positive and sero negative participants received IV dose of inebilizumab 300 mg on Day 1 and Day 15 of RCP. The participants who entered OLP received IV inebilizumab 300 mg on Day 1 and matching placebo on Day 15, followed by a single IV dose of inebilizumab 300 mg every 6 months until maximum of 3 years after the last participant enters the OLP. Participants had choice to enter in the SFP at any point during RCP or OLP and were free to pursue other treatment options otherwise prohibited during the RCP and OLP. Participants continued in the SFP for 12 months from last dose of study drug.
Period: Randomized-controlled Period (RCP)
Arm/Group | Placebo/Inebilizumab | Inebilizumab/Inebilizumab
Started | 56 | 175
Treated | 56 | 174
Completed | 54 | 169
Not Completed | 2 | 6
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Participants randomized, but not treated | 0 | 1
Not completed — Other | 1 | 2
Period: Open-label Period (OLP)
Arm/Group | Placebo/Inebilizumab | Inebilizumab/Inebilizumab
Started | 51 (3 participants completed RCP but did not roll over to OLP.) | 165 (4 participants completed RCP but did not roll over to OLP.)
Completed | 43 | 131
Not Completed | 8 | 34
Not completed — Adverse Event | 1 | 2
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 14
Not completed — Other | 6 | 15

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) population included all participants who were randomized, received any study drug, and grouped according to their randomized treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Inebilizumab | Inebilizumab/Inebilizumab | Total
Number analyzed (Participants) | 56 | 174 | 230
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.6 (13.9) | 43.0 (11.6) | 42.9 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 159 | 209
  Male | 6 | 15 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 28 | 43
  Not Hispanic or Latino | 41 | 146 | 187
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 14 | 19
  Asian | 8 | 39 | 47
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 15 | 20
  White | 28 | 92 | 120
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 10 | 13 | 23

OUTCOME MEASURES:

1. Primary Outcome: Time to Adjudication Committee (AC)-Determined Neuromyelitis Optica Spectrum Disorder (NMOSD) Attack During RCP
Description: The NMOSD attack is defined as the presence of new or worsening symptom(s) related to NMOSD that meet at least one of the 18 protocol-defined attack criteria. These criteria were developed in conjunction with a panel of disease experts and with Food and Drug Administration input, and were intended to be clinically meaningful, objective, quantifiable, and able to be used worldwide. Only attacks positively adjudicated by the AC were used for the primary analysis.
Time Frame: Day 1 (Baseline) through Day 197
Population: The ITT population included all participants who were randomized, received any study drug, and grouped according to their randomized treatment.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo/Inebilizumab | Inebilizumab/Inebilizumab
Number analyzed (Participants) | 56 | 174
Days | NA [142.0 to NA] — Median and upper level of 95% Confidence Interval (CI) are not reported as there were insufficient events to determine the median. | NA [NA to NA] — Median and 95% CI are not reported as there were insufficient events to determine the median.
Statistical Analysis 1: Comparison: Placebo/Inebilizumab vs Inebilizumab/Inebilizumab; Test type: Superiority; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.272, 95% CI 2-sided [0.1496 to 0.4961]

2. Secondary Outcome: Percentage of Participants With Worsening in Expanded Disability Severity Scale (EDSS) Score From Baseline to the Last Visit of RCP
Description: EDSS and its associated functional system (FS) score provide a system for quantifying disability and monitoring changes in the level of disability over time. EDSS is a scale for assessing neurologic impairment in multiple sclerosis (MS). It consists of 7 FS (visual FS, brainstem FS, pyramidal FS, cerebellar FS, sensory FS, bowel and bladder FS, and cerebral FS) which are used to derive EDSS score ranging from 0 (normal neurological exam) to 10 (death from MS). A negative change from baseline indicates improvement. A participant was considered to have a worsening in overall EDSS score of at least 2 if baseline EDSS score was 0, or at least 1 point if baseline EDSS score is 1 to 5, or at least 0.5 point if baseline EDSS score is 5.5 or more.
Time Frame: Day 1 (Baseline) through Day 197
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo/Inebilizumab | Inebilizumab/Inebilizumab
Number analyzed (Participants) | 56 | 174
Percentage of Participants | 33.9 | 14.9
Statistical Analysis 1: Comparison: Placebo/Inebilizumab vs Inebilizumab/Inebilizumab; Test type: Superiority; p = 0.0033, Regression, Logistic; Odds Ratio (OR) = 0.352, 95% CI 2-sided [0.1755 to 0.7059]

3. Secondary Outcome: Change From Baseline in Low-Contrast Visual Acuity Binocular Score to the Last Visit of RCP
Description: Low-contrast visual acuity test is used to determine the number of letters that can be read on a standardized low-contrast Landolt C Broken Rings Chart held at a distance of 3 meters. Binocular score is the number of letters read correctly on an eye chart using both eyes simultaneously. The total score ranges from 0-70. Higher score indicates better vision.
Time Frame: Day 1 (Baseline) through Day 197
Population: The ITT population included all participants who were randomized, received any study drug, and grouped according to their randomized treatment. Participants with low contrast visual acuity binocular score were analyzed for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo/Inebilizumab | Inebilizumab/Inebilizumab
Number analyzed (Participants) | 56 | 171
Score on scale | 1.442 (1.217) | 1.576 (0.935)
Statistical Analysis 1: Comparison: Placebo/Inebilizumab vs Inebilizumab/Inebilizumab; Test type: Superiority; p = 0.9026, ANCOVA; Mean Difference (Net) = 0.134, 95% CI 2-sided [-2.0254 to 2.2941], Standard Error of Mean 1.096

4. Secondary Outcome: Cumulative Number of Active Magnetic Resonance Imaging (MRI) Lesions During RCP
Description: The number of new gadolinium-enhancing lesions and new or enlarging T2 lesions were measured by MRI of the brain, optic nerve, and spinal cord.
Time Frame: From Screening (Day -28) to Day 197
Population: The ITT population included all participants who were randomized, received any study drug, and grouped according to their randomized treatment. Participants with observed MRI lesions were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: Number of lesions
Arm/Group | Placebo/Inebilizumab | Inebilizumab/Inebilizumab
Number analyzed (Participants) | 32 | 79
Number of lesions | 2.3 (1.3) | 1.6 (1.0)
Statistical Analysis 1: Comparison: Placebo/Inebilizumab vs Inebilizumab/Inebilizumab; Test type: Superiority; p = 0.0034, Negative Binomial Regression; Rate Ratio = 0.566, 95% CI 2-sided [0.3866 to 0.8279]

5. Secondary Outcome: Number of NMOSD-related In-patient Hospitalizations During RCP
Description: Participants with relapsing NMOSD have recurrent attacks that can be severe and result in blindness, paralysis, and even death and consequently, such attacks frequently result in in-patient hospitalizations. In-patient hospitalization is defined as a stay in hospital that goes beyond midnight of the first day of admission.
Time Frame: Day 1 (Baseline) through Day 197
Population: The ITT population included all participants who were randomized, received any study drug, and grouped according to their randomized treatment. Participants with in-patient hospitalization were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: Number of In-patient Hospitalizations
Arm/Group | Placebo/Inebilizumab | Inebilizumab/Inebilizumab
Number analyzed (Participants) | 8 | 11
Number of In-patient Hospitalizations | 1.4 (0.7) | 1.0 (0)
Statistical Analysis 1: Comparison: Placebo/Inebilizumab vs Inebilizumab/Inebilizumab; Test type: Superiority; p = 0.0146, Negative Binomial Regression; Rate Ratio = 0.317, 95% CI 2-sided [0.1257 to 0.7972]

6. Secondary Outcome: Annualized AC-determined NMOSD Attack Rate During Any Exposure to Inebilizumab
Description: Annualized attack rate is defined as total number of AC-determined attacks divided by total person years. Total person-years is calculated as the sum of the person-years for individual participant. Person-year for individual participant = (Date of last day before safety follow-up period - first inebilizumab dose date +1)/365.25. Annualized AC-determined NMOSD attack rate during any exposure to inebilizumab (in RCP and OLP) is reported.
Time Frame: For participants randomized to inebilizumab: Day 1 of RCP through end of OLP (approximately 3.5 years); and for participants randomized to placebo: Day 1 of OLP through the end of OLP (approximately 3 years)
Population: Any inebilizumab population included all participants who received at least one dose of inebilizumab either in the RCP or OLP.
Measure: Number; unit: Annualized attack rate
Groups:
- Any Inebilizumab: AQP4-IgG sero positive and sero negative participants received IV dose of inebilizumab 300 mg on Day 1 and Day 15 in RCP or IV inebilizumab 300 mg on both Day 1 and Day 15 in OLP ; followed by a single IV dose of inebilizumab 300 mg every 6 months until maximum of 3 years after the last participant enters the OLP.
Arm/Group | Any Inebilizumab
Number analyzed (Participants) | 225
Annualized attack rate | 0.086

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs) During RCP
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event is any AE that resulted in death, life threatening, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, is a congenital anomaly/birth defect in offspring of a study participant, is an important medical event that may jeopardize the participant or may require medical intervention. TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug during the RCP.
Time Frame: Day 1 (Baseline) through Day 197
Population: As-treated population included all participants who received any dose of study drug and analyzed according to the treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Inebilizumab | Inebilizumab/Inebilizumab
Number analyzed (Participants) | 56 | 174
Participants
  TEAEs | 41 | 127
  TESAEs | 6 | 9

8. Secondary Outcome: Number of Participants With TEAEs and TESAEs During OLP
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event is any AE that resulted in death, life threatening, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, is a congenital anomaly/birth defect in offspring of a study participant, is an important medical event that may jeopardize the participant or may require medical intervention. TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug during the OLP.
Time Frame: Day 198 through end of OLP period (maximum of 3 years after the last participant entered, until regulatory approval or study discontinuation, whichever occurs first) (approximately 3 years)
Population: Open-label population included all participants who received at least one dose of inebilizumab during OLP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Inebilizumab | Inebilizumab/Inebilizumab
Number analyzed (Participants) | 51 | 165
Participants
  TEAEs | 45 | 144
  TESAEs | 19 | 22

9. Secondary Outcome: Number of Participants With TEAEs and TESAEs During SFP (Open-label Population)
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event is any AE that resulted in death, life threatening, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, is a congenital anomaly/birth defect in offspring of a study participant, is an important medical event that may jeopardize the participant or may require medical intervention. TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug during the OLP. Participant who prematurely discontinued from the RCP or OLP entered in the SFP.
Time Frame: Every 3 months for a total of 1 year after the last dose of study drug (approximately 3 years)
Population: Open-label population included all participants who received at least one dose of inebilizumab during OLP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Inebilizumab | Inebilizumab/Inebilizumab
Number analyzed (Participants) | 51 | 165
Participants
  TEAEs | 3 | 5
  TESAEs | 2 | 1

10. Secondary Outcome: Number of Participants With TEAEs and TESAEs During SFP (Non-OLP Population)
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event is any AE that resulted in death, life threatening, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, is a congenital anomaly/birth defect in offspring of a study participant, is an important medical event that may jeopardize the participant or may require medical intervention. TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug during the OLP. The SFP started when a participant prematurely discontinues from the RCP or OLP.
Time Frame: Every 3 months for a total of 1 year after the last dose of study drug (approximately 3 years)
Population: Non-OLP population included all participants who received any dose of study drug, analyzed according to the treatment received in RCP, but did not roll over to OLP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Inebilizumab | Inebilizumab/Inebilizumab
Number analyzed (Participants) | 5 | 9
Participants
  TEAEs | 2 | 3
  TESAEs | 1 | 1

11. Secondary Outcome: Number of Participants With at Least a 2-Grade Shift From Baseline to Worst Toxicity Grade in Hematology and Chemistry During RCP
Description: Number of participants with at least a 2-grade shift from baseline to worst toxicity grade in hematology and chemistry during RCP is reported.
Time Frame: Day 1 (Baseline) through Day 197
Population: As-treated population included all participants who received any dose of study drug and analyzed according to the treatment received. 'Number of Participants analyzed' signifies participants who were analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Inebilizumab | Inebilizumab/Inebilizumab
Number analyzed (Participants) | 56 | 173
Participants
  Hemoglobin (decreased) | 0 | 2
  Leukocytes (decreased) | 1 | 11
  Lymphocytes (decreased) | 5 | 35
  Lymphocytes (increased) | 4 | 1
  Neutrophils (decreased) | 0 | 10
  Alanine Aminotransferase (increased) | 1 | 4
  Aspartate Aminotransferase (increased) | 2 | 1
  Bilirubin (increased) | 2 | 1
  Cholesterol (increased) | 2 | 5
  Creatinine (increased) | 1 | 5
  Gamma glutamyl transferase (increased) | 1 | 6
  Glucose (decreased) | 1 | 1
  Glucose (increased) | 5 | 1
  Potassium (decreased) | 0 | 1
  Sodium (decreased) | 1 | 2
  Triglycerides (increased) | 2 | 7

12. Secondary Outcome: Number of Participants With at Least a 2-Grade Shift From Baseline to Worst Toxicity Grade in Hematology and Chemistry During OLP
Description: Number of participants with at least a 2-grade shift from baseline to worst toxicity grade in hematology and chemistry during OLP is reported.
Time Frame: Day 198 through end of OLP (maximum of 3 years after the last participant enters, until regulatory approval or study discontinuation, whichever occurs first) (approximately 3 years)
Population: Open-label population included all participants who received at least one dose of study drug during OLP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Inebilizumab | Inebilizumab/Inebilizumab
Number analyzed (Participants) | 51 | 165
Participants
  Hemoglobin (decreased) | 2 | 6
  Leukocytes (decreased) | 1 | 12
  Lymphocytes (decreased) | 9 | 21
  Lymphocytes (increased) | 1 | 4
  Neutrophils (decreased) | 1 | 16
  Alanine aminotransferase (increased) | 4 | 2
  Albumin (decreased) | 0 | 3
  Alkaline phosphatase (increased) | 1 | 1
  Aspartate aminotransferase (increased) | 2 | 3
  Cholesterol (increased) | 1 | 5
  Creatinine (increased) | 3 | 7
  Gamma glutamyl transferase (increased) | 1 | 10
  Glucose (decreased) | 0 | 3
  Glucose (increased) | 5 | 5
  Potassium (decreased) | 0 | 1
  Potassium (increased) | 1 | 2
  Sodium (decreased) | 2 | 1
  Triglycerides (increased) | 4 | 6
  Urate (increased) | 1 | 1
  Hemoglobin (increased) | 0 | 1
  Bilirubin | 2 | 0

13. Secondary Outcome: Time to Maximum Serum Concentration (Tmax) of Inebilizumab (During RCP)
Description: Time to maximum serum concentration of inebilizumab during RCP is reported.
Time Frame: Dose 1 (Pre and post dose on Day 1 and Day 8); and Dose 2 (pre and post dose on Day 15; and Days 29, 57, 85, 113, 155, and 197)
Population: The ITT population included all participants who were randomized, received any study drug, and grouped according to their randomized treatment. 'Number analyzed' signifies participants who had adequate pharmacokinetic sample of inebilizumab per the specified dose levels (Dose 1 and Dose 2).
Measure: Median (Full Range); unit: Days
Arm/Group | Inebilizumab/Inebilizumab
Number analyzed (Participants) | 173
Days
  Dose 1 | 0.07 [0.07 to 7.00]
  Dose 2: number analyzed (Participants) | 168
  Dose 2 | 0.07 [0.07 to 14.00]

14. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Inebilizumab (During RCP)
Description: Maximum observed serum concentration of inebilizumab during RCP is reported.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Inebilizumab/Inebilizumab
Number analyzed (Participants) | 173
μg/mL
  Dose 1 | 97.7 (37.4)
  Dose 2: number analyzed (Participants) | 168
  Dose 2 | 108 (45.4)

15. Secondary Outcome: Area Under the Serum Concentration Time Curve of the Dosing Interval (AUC0-14d) of Inebilizumab (During RCP)
Description: Area under the serum concentration time curve of the dosing interval (AUC0-14d) of inebilizumab during RCP is reported.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*d/mL
Arm/Group | Inebilizumab/Inebilizumab
Number analyzed (Participants) | 167
μg*d/mL
  Dose 1 | 667 (31.3)
  Dose 2: number analyzed (Participants) | 164
  Dose 2 | 967 (39.6)

16. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADA) Titer to Inebilizumab (During RCP)
Description: Number of participants with positive ADA titer to inebilizumab during RCP is reported.
Time Frame: Pre and post dose on Day 1; and on Days 29, 85, and 197
Population: The ITT population included all participants who were randomized, received any study drug, and grouped according to their randomized treatment. 'Number analyzed' signifies the number of participants who had adequate ADA samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Inebilizumab | Inebilizumab/Inebilizumab
Number analyzed (Participants) | 56 | 174
Participants
  ADA positive at anytime including baseline (BL) | 8 | 17
  ADA positive at BL; not detected post-BL: number analyzed (Participants) | 56 | 171
  ADA positive at BL; not detected post-BL | 0 | 5
  ADA positive post-BL; positive at BL: number analyzed (Participants) | 56 | 171
  ADA positive post-BL; positive at BL | 4 | 7
  ADA positive post-BL; not detected at BL: number analyzed (Participants) | 56 | 171
  ADA positive post-BL; not detected at BL | 4 | 5

17. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADA) Titer to Inebilizumab (During OLP)
Description: Number of participants with positive ADA titer to inebilizumab in OLP is reported.
Time Frame: Pre and post dose on Day 1; and on Days 92, 183, 274, and then every 6 months (maximum of 3 years after the last participant enters, until regulatory approval or study discontinuation, whichever occurs first) (approximately 3 years)
Population: Open-label population included all participants who received at least one dose of inebilizumab during OLP. 'Number analyzed' signifies the number of participants who had adequate ADA samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Inebilizumab | Inebilizumab/Inebilizumab
Number analyzed (Participants) | 51 | 165
Participants
  ADA positive at any time including baseline (BL) | 9 | 22
  ADA positive at BL; not detected post-BL: number analyzed (Participants) | 51 | 162
  ADA positive at BL; not detected post-BL | 0 | 5
  ADA positive post-BL and positive at BL: number analyzed (Participants) | 51 | 162
  ADA positive post-BL and positive at BL | 4 | 7
  ADA positive post-BL; not detected at BL: number analyzed (Participants) | 51 | 162
  ADA positive post-BL; not detected at BL | 5 | 10

ADVERSE EVENTS:
Time Frame: From Day 1 through the end of study (approximately 5 years 10 months)
Description: Adverse events are reported for all 3 study periods combined (RCP, OLP, and SFP).
Arm/Group | Placebo/Inebilizumab | Inebilizumab/Inebilizumab
All-Cause Mortality (participants affected / at risk) | 1/56 | 2/174
Serious Adverse Events (participants affected / at risk) | 24/56 | 28/174
Other Adverse Events (participants affected / at risk) | 48/56 | 138/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Inebilizumab (N=56) | Inebilizumab/Inebilizumab (N=174)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Renal abscess (Infections and infestations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Optic neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral nerve palsy (Nervous system disorders) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Steroid withdrawal syndrome (Endocrine disorders) | 0 (0) | 1 (1)
Blindness unilateral (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (2)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Central nervous system infection (Infections and infestations) | 0 (0) | 1 (1)
Chorioretinitis (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis a (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0)
Neuroborreliosis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 3 (5)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Progressive multifocal leukoencephalopat (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis chronic (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 7 (11) | 3 (3)
Burns third degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Lumbosacral radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Myelitis transverse (Nervous system disorders) | 0 (0) | 1 (1)
Neuromyelitis optica spectrum disorder (Nervous system disorders) | 2 (2) | 3 (3)
Post cardiac arrest syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Unresponsive to stimuli (Nervous system disorders) | 1 (2) | 0 (0)
Uraemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Drug reaction with eosinophilia and syst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Inebilizumab (N=56) | Inebilizumab/Inebilizumab (N=174)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 11 (12)
Dry eye (Eye disorders) | 6 (6) | 4 (4)
Eye pain (Eye disorders) | 5 (5) | 8 (27)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 3 (3)
Constipation (Gastrointestinal disorders) | 7 (7) | 9 (13)
Diarrhoea (Gastrointestinal disorders) | 8 (10) | 15 (19)
Gastritis (Gastrointestinal disorders) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 9 (9) | 15 (31)
Vomiting (Gastrointestinal disorders) | 6 (8) | 9 (11)
Fatigue (General disorders) | 3 (3) | 12 (16)
Influenza like illness (General disorders) | 4 (6) | 3 (6)
Pyrexia (General disorders) | 5 (12) | 9 (12)
Bronchitis (Infections and infestations) | 5 (6) | 12 (13)
Conjunctivitis (Infections and infestations) | 3 (5) | 5 (6)
Influenza (Infections and infestations) | 4 (10) | 17 (20)
Nasopharyngitis (Infections and infestations) | 11 (17) | 38 (69)
Oral herpes (Infections and infestations) | 4 (8) | 5 (6)
Rhinitis (Infections and infestations) | 2 (3) | 9 (10)
Upper respiratory tract infection (Infections and infestations) | 10 (15) | 28 (51)
Urinary tract infection (Infections and infestations) | 20 (54) | 40 (77)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 11 (18)
Infusion related reaction (Injury, poisoning and procedural complications) | 9 (16) | 22 (47)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (14) | 28 (37)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (6) | 5 (8)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (6) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (14) | 11 (20)
Dizziness (Nervous system disorders) | 3 (3) | 7 (7)
Headache (Nervous system disorders) | 13 (16) | 31 (82)
Hypoaesthesia (Nervous system disorders) | 2 (3) | 12 (24)
Paraesthesia (Nervous system disorders) | 2 (2) | 12 (15)
Depression (Psychiatric disorders) | 6 (6) | 8 (8)
Insomnia (Psychiatric disorders) | 6 (6) | 10 (10)
Micturition urgency (Renal and urinary disorders) | 3 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (15) | 17 (20)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5)
Eczema (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 4 (6) | 7 (11)
Hypertension (Vascular disorders) | 3 (4) | 5 (11)
Hypotension (Vascular disorders) | 4 (4) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 24 (38)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 3 (5)

LIMITATIONS AND CAVEATS:
In the safety follow-up period (SFP), only 1 participant from 'Placebo/Inebilizumab' arm rolled over to SFP and no participant from 'Inebilizumab /Inebilizumab' arm rolled over to SFP. For EudraCT result posting, a study period with any one of the arm with zero participants started is not acceptable (EudraCT limitation). Therefore, not included SFP in 'Participant Flow' section to keep the data consistent across registry portals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Viela Bio has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it is understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multicentre publication.

DOCUMENTS (2):
  • Study Protocol (2018-10-11): https://cdn.clinicaltrials.gov/large-docs/70/NCT02200770/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/70/NCT02200770/SAP_001.pdf